CLINICAL TRIAL: NCT07103733
Title: Percutaneous or Surgical Repair In Mitral Prolapse And Regurgitation for ≥60 Year-olds (PRIMARY) Ancillary Substudy
Brief Title: PRIMARY Ancillary Substudy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Annetine Gelijns (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Annetine Gelijns, Department Chair, Department of Population Health Science & Policy Edmond A. Guggenheim Professor of Health Policy Co-Director, InCHOIR, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GCO 08-1078 ANC; 5U01HL088942-17 (NIH)
Record Dates: First submitted 2025-07-22; First posted 2025-08-05 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Mitral Valve Prolapse; Left Ventricular Fibrosis; Ventricular Arrhythmias
Keywords: Mitral valve repair (MVr); Transcatheter-edge-to-edge-repair (TEER); Cardiac magnetic resonance imaging (CMR); ZioPatch monitoring; Heart biopsy
MeSH Terms: conditions — Mitral Valve Prolapse

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The PRIMARY trial is an open-label trial. As in the parent trial, clinical investigators, and coordinators, however, will be blinded to all overall outcome data in the ancillary study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Mitral valve repair (Active Comparator): Mitral surgery will be conducted using general anesthesia and cardiopulmonary bypass. Mitral surgery may be performed via a sternotomy or a right thoracotomy approach with or without robotic assistance.
  Interventions: Procedure: Cardiac Magnetic Resonance Imaging; Device: ZioPatch Monitoring; Procedure: Myocardial Tissue Biopsy
- Transcatheter edge-to-edge repair (Active Comparator): Patients will be treated with a commercially-approved edge-to-edge mitral repair device.
  Interventions: Procedure: Cardiac Magnetic Resonance Imaging; Device: ZioPatch Monitoring

INTERVENTIONS:
Procedure: Cardiac Magnetic Resonance Imaging — Non-invasive imaging test that uses powerful magnets and radio waves to create detailed pictures of the heart without using radiation.
  Other Names: CMR
Device: ZioPatch Monitoring — ZioPatch is a small, wearable heart monitor that sticks to the chest and records the heart's electrical activity continuously for up to 14 days. It helps doctors detect irregular heart rhythms (arrhythmias) without the need for bulky wires or equipment.
  Other Names: iRhythm Monitoring
Procedure: Myocardial Tissue Biopsy — During the MVr procedure, surgeons will biopsy approximately 50 μg of tissue from the endocardial and subendocardial myocardium in the inferobasilar and control areas using a surgical rongeur.
  Other Names: Heart Bioplsy
  Arms: Mitral valve repair

SUMMARY:
The PRIMARY trial (NCT05051033), which compares mitral valve repair (MVr) to transcatheter-edge-to-edge-repair (TEER), offers a platform for conducting mechanistic studies to develop early insights into the pathophysiological processes by which mitral valve prolapse (MVP) can impact left ventricular (LV) myocardial structure and function, and, thereby, predispose to arrhythmias and sudden death. Such insights are key to identifying interventions to reduce the long-term sequelae of heart failure (HF) and arrhythmias, as well as delineate optimal therapeutic approaches for different patient sub-groups.

DETAILED DESCRIPTION:
This is an ancillary study of a multicenter randomized clinical trial comparing MVr to TEER for degenerative mitral regurgitation (MR) involving up to 250 patients from the parent trial. All patients will receive rhythm monitoring, up to 200 patients will receive pre/post intervention CMR, all patients in the parent trial will undergo a transthoracic echocardiogram (TTE) (as part of the randomized controlled trial (RCT)), and 60 surgical patients will undergo tissue biopsies. The study is being conducted in highly experienced clinical centers in the U.S., Canada, Germany, the U.K. and Spain. The estimated enrollment period is 12-18 months. Outcomes will be measured from baseline to 12 months after randomization.

This mechanistic ancillary study has the following aims:

1. To compare the impact of MVr and TEER on disordered ventricular biomechanics and myocardial fibrosis that predispose to ventricular arrhythmias, using speckle tracking strain echocardiography, cardiac magnetic resonance imaging (CMR), and rhythm monitoring pre- and post-mitral valve (MV) intervention. The research team hypothesize's that a treatment strategy that more effectively and durably reduces MVP and MR will lead to improved ventricular mechanics, limit progression of myocardial fibrosis and decrease the burden of ventricular arrhythmias and HF.
2. To compare the impact of MVr and TEER on recurrent/residual MR, LV and left atrial (LA) reverse remodeling with baseline and 1-year post-intervention CMR, and to use quantitative CMR myocardial tissue phenotyping as a predictor of response to MVr and TEER.
3. To construct functional pre-operative CMR fingerprints that recapitulate the mechanical state of the heart to develop individualized computational models, which will be altered in silico based on the proposed treatment plan, to predict patients' response to therapy. These results will be validated against post-operative outcome data to test the validity of this approach for predicting treatment response.
4. To explore the relationships among gene products, structural variables, and post-operative clinical outcomes, including reverse remodeling, using tissue obtained at surgery from ventricular myocardium.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all eligibility criteria and are randomized in the parent PRIMARY trial.
* For the ancillary biospecimen study, patients who are randomized to MVr in the parent trial.

Exclusion Criteria:

* Severe claustrophobia not controlled with sedation.
* Prior adverse reaction to gadolinium administration.
* Patients with an implantable subcutaneous cardioverter defibrillator and/or cardiac resynchronization therapy device with defibrillator may be excluded as they typically produce substantial artifacts on cardiac MRI making assessment very challenging.
* Known allergic reaction to adhesives or hydrogels or with family history of adhesive skin allergies (for patients undergoing rhythm monitoring).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Presence of Myocardial Fibrosis | 1 year post index procedure.
  Myocardial fibrosis is the buildup of excess fibrous connective tissue in the heart muscle often resulting from chronic injury or stress. It can impair the heart's ability to contract and relax properly leading to reduced cardiac function.
Presence of Ventricular Arrythmia | 1 year post index procedure.
  A ventricular arrhythmia is an abnormal heart rhythm that starts in the lower chambers of the heart (the ventricles). It can cause the heart to beat too fast, which may reduce blood flow to the body and, in some cases, be life-threatening.
Proteomics | 1 year post index procedure.
  Proteomics is the large-scale study of proteins, which are essential molecules that carry out most functions in the body. By analyzing proteins in tissues or fluids, scientists can better understand diseases, identify biomarkers, and discover new treatment targets.

SECONDARY OUTCOMES:
Computational and Predictive Models of Treatment Outcome | 1 year post index procedure.
  specific treatment. These tools help doctors make more personalized and effective care decisions based on patterns found in large sets of medical information.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Chikwe, MD, Study Director — Cedars-Sinai; Martin Leon, MD, Study Director — Columbia University
Locations (25):
- United States (16):
  - Keck Hospital of the University of Southern California, Los Angeles, California
  - Cedars-Sinai, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Piedmont Heart Institute, Atlanta, Georgia
  - Maine Medical Center, Portland, Maine
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Saint Luke's Hospital of Kansas City/MidAmerica Heart and Lung Surgeons, Kansas City, Missouri
  - Weill Cornell Medicine/ New York-Presbyterian Hospital, New York, New York
  - Northwell--Lenox Hill, North Shore, South Shore, Staten Island University Hospital, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Virginia Medical Center, Charlottesville, Virginia
  - West Virginia University Hospital, Morgantown, West Virginia
- Germany (2):
  - Deutsches Herzzentrum der Charité, Berlin
  - Herzzentrum Leipzig, Leipzig
- United Kingdom (7):
  - Royal Papworth Hospital NHS Foundation Trust, Trumpington, Cambridge
  - The Leeds Teaching Hospitals NHS Trust, Leeds, England
  - Barts Health NHS Trust, Whitechapel, London
  - Manchester University NHS Foundation Trust, Oxford, Manchester
  - South Tees Hospitals NHS Foundation Trust, Marton-in-Cleveland, Middlesbrough
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - University Hospitals Sussex NHS Foundation Trust, Worthing, West Sussex

IPD SHARING:
Plan to Share IPD: No
Data shared will be in aggregate.

REFERENCES:
- See also: PRIMARY Trial — https://clinicaltrials.gov/study/NCT05051033